CLINICAL TRIAL: NCT00424476
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 52-Wk Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Belimumab in Subjects With Systemic Lupus Erythematosus (SLE)
Acronym: BLISS-52
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGS1006-C1057; BLISS-52 (Other: Human Genome Sciences Inc.); 110752 (Other: GSK)
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmune Diseases; Lupus; SLE; Systemic Lupus Erythematosus; Belimumab; Antibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Belimumab 1 mg/kg (Experimental): Belimumab 1 mg/kg
  Interventions: Drug: Belimumab 1 mg/kg
- Belimumab 10 mg/kg (Experimental): Belimumab 10 mg/kg
  Interventions: Drug: Belimumab 10 mg/kg

INTERVENTIONS:
Drug: Placebo — Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through Week 48.
  Arms: Placebo
Drug: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV plus standard therapy on Days 0, 14, 28, and every 28 days thereafter through Week 48.
  Other Names: BENLYSTA™ (formerly LymphoStat-B™)
  Arms: Belimumab 1 mg/kg
Drug: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV plus standard therapy on Days 0, 14, 28, and every 28 days thereafter through Week 48.
  Other Names: BENLYSTA™ (formerly LymphoStat-B™)
  Arms: Belimumab 10 mg/kg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, and impact on quality of life of two different doses of belimumab administered in addition to standard therapy in subjects with active, autoantibody-positive systemic lupus erythematosus (SLE) disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by ACR criteria.
* Active SLE disease.
* Autoantibody-positive.
* On stable SLE treatment regimen.

Key Exclusion Criteria:

* Pregnant or nursing
* Have received treatment with any B cell targeted therapy.
* Have received treatment with a biological investigational agent in the past year.
* Have received IV cyclophosphamide within 180 days of Day 0.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have required management of acute or chronic infections within the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test positive at screening for HIV, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — Human Genome Sciences Inc.
Locations (92):
- Argentina (11):
  - OMI, Organización Médica de Investigación, Buenos Aires
  - CIER, Centro de Investigaciones en Enfermedades Reumáticas, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital General de Agudos Carlos G. Durand, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Hospital Sirio Libanes, Buenos Aires
  - Atencion Integral en Reumatologia, Buenos Aires
  - Instituto de Investigaciones Medicas, Buenos Aires
  - Hospital Interzonal General San Martín, La Plata
  - CAICI, Instituto Centralizado de Asistencia e Investigación Clínica Integral, Rosario
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Australia (4):
  - Repatriation Hospital, Daw Park
  - Emeritus Research, Cabrini Hospital, Melbourne
  - Monash Medical Centre, Melbourne
  - Royal Perth Hospital, Shenton Park
- Brazil (12):
  - Hospital de Clínicas - UNICAMP, Campinas
  - Hospital das Clínicas - Universidade do Paraná, Curitiba
  - Hospital de Clínicas - Universidade Federal de Pernambuco, Fortaleza
  - Hospital Geral de Goiânia, Goiânia
  - Hospital Universitário - Universidade Federal de Juiz de Fora, Juiz de Fora
  - Hospital São Lucas da PUC-RS, Porto Alegre
  - Hospital Universitário Pedro Ernesto - UERJ, Rio de Janeiro
  - Hospital Unversitario Clementino Fraga Filho UFRJ, Rio de Janeiro
  - Hospital Santa Izabel, Salvador
  - Hospital Abreu Sodré, São Paulo
  - Hospital do Servidor Público Estadual de São Paulo - Francisco Morato de Oliveira, São Paulo
  - Hospital Heliópolis, São Paulo
- Chile (4):
  - Hospital Dr. Sotero del Rio, Santiago
  - Pontificia Universidad Católica de Chile, Santiago
  - Clínica Dávila, Santiago
  - Hospital Dr. Gustavo Fricke, Viña del Mar
- Colombia (9):
  - Office of Dr. Guzman, Bogota, Cundinamarca
  - Fundación Oftalmologica de Santander Clinica Carlos Ardila Lulle, Bucaramanga, Santander Department
  - Centro de Reumatologia y Ortopedia, Barranquilla
  - Centrode de Investigaciones en Reumatologia Especialidades Medicas (CIREEH), Bogotá
  - Fundación Instituto de Reumatología Fernando Chalem, Bogotá
  - Riesgo de Fracturas, Bogotá
  - SERVIMED, Bucaramanga
  - Corporación para Investigaciones Biológicas (CIB), Medellín
  - Office of Dr. Jose Molina, Medellín
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Rheumatology Assessment and Treatment Center, Pok Oi Hospital, Shatin
  - Tuen Mun Hospital, Tuenmen
- India (7):
  - St. John's Medical College Hospital, Bangalore
  - Krishna Institute of Medical Sciences, Hyderabaad
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Apollo Hospitals, Hyderabad
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow
  - King Edward Memorial (K.E.M.) Hospital, Mumbai
  - Kerala Institute of Medical Sciences, Trivandrum
- Peru (4):
  - Hospital Nacional Alberto Sabogal Sologuren ESSALUD, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen ESSALUD, Lima
  - Clinica Ricardo Palma Anexo 9 - Javier Prado Este, Lima
  - Instituto de Ginecología y Reproducción, Lima
- Philippines (6):
  - Chong Hua Hospital, Cebu City
  - Davao Medical Center, Davao City
  - University of Perpetual Help -Rizal, Las Piñas
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
- Romania (5):
  - Spitalul Clinic Sf Maria, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul de Urgenta al Ministerului Administratiei si Internelor Prof. Dr. Dimitrie Gerota, Bucharest
  - Spitalul Clinic Dr. Ion Cantacuzino, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
- Russia (6):
  - State Institution Scientific Research Institute of Rheumatology, Moscow
  - St. Petersburg City Hospital (Rheumatology Center), Saint Petersburg
  - Academy of Post-Graduated Education, Saint Petersburg
  - St.-Petersburg Region Clinical Hospital, Saint Petersburg
  - Soloviev's City Clinical Hospital,, Yaroslavl
  - City Healthcare Institution Municipal Hospital NPZ,, Yaroslavl
- South Korea (10):
  - Kyungpook National Univesity Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Inha University Hospital, Inchon
  - Dong-A University Hospital 3-1 (Dept. Rhuematology), Pusan
  - Pusan National University Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - The Hospital for Rheumatic Diseases, Hanyang University Hospital, Seoul
  - Catholic Universtigy of Korea, Kangnam St. Mary's Hospital, Seoul
  - Catholic University, Yoido St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (11):
  - Buddhist Tzu Chi General Hospital, Dalin, Chiayi City
  - Buddhist Tzu Chi General Hospital - Hualien, Haulien
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaosiung, Kaosiung
  - Chang Gung Memorial Hospital-Keelung, Keelung
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linko, Tau-Yuan County

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Botto J, Cetrez N, Nikolopoulos D, Regardt M, Heintz E, Lindblom J, Parodis I. Predicting EQ-5D full health state in systemic lupus erythematosus using machine learning algorithms. Rheumatol Adv Pract. 2025 Apr 18;9(2):rkaf032. doi: 10.1093/rap/rkaf032. eCollection 2025. PMID 40256631
- [Derived] Nikolopoulos D, Cetrez N, Lindblom J, Parodis I. Neuropsychiatric involvement in systemic lupus erythematosus contributes to organ damage beyond the nervous system: a post-hoc analysis of 5 phase III randomized clinical trials. Rheumatol Int. 2024 Sep;44(9):1679-1689. doi: 10.1007/s00296-024-05667-5. Epub 2024 Aug 8. PMID 39115551
- [Derived] Jesus D, Henriques C, Matos A, Doria A, Ines LS. Systemic Lupus Erythematosus Disease Activity Score Remission and Low Disease Activity States Discriminate Drug From Placebo and Better Health-Related Quality of Life. Arthritis Care Res (Hoboken). 2024 Jun;76(6):788-795. doi: 10.1002/acr.25305. Epub 2024 Feb 29. PMID 38258369
- [Derived] Jagerback S, Gomez A, Parodis I. Predictors of renal flares in systemic lupus erythematosus: a post-hoc analysis of four phase III clinical trials of belimumab. Rheumatology (Oxford). 2025 Feb 1;64(2):623-631. doi: 10.1093/rheumatology/keae023. PMID 38216728
- [Derived] Emamikia S, Oon S, Gomez A, Lindblom J, Borg A, Enman Y, Morand E, Grannas D, van Vollenhoven RF, Nikpour M, Parodis I. Impact of remission and low disease activity on health-related quality of life in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2022 Nov 28;61(12):4752-4762. doi: 10.1093/rheumatology/keac185. PMID 35302581
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Derived] Rendas-Baum R, Baranwal N, Joshi AV, Park J, Kosinski M. Psychometric properties of FACIT-Fatigue in systemic lupus erythematosus: a pooled analysis of three phase 3 randomised, double-blind, parallel-group controlled studies (BLISS-SC, BLISS-52, BLISS-76). J Patient Rep Outcomes. 2021 Apr 8;5(1):33. doi: 10.1186/s41687-021-00298-x. PMID 33830377
- [Derived] Maslen T, Bruce IN, D'Cruz D, Ianosev M, Bass DL, Wilkinson C, Roth DA. Efficacy of belimumab in two serologically distinct high disease activity subgroups of patients with systemic lupus erythematosus: post-hoc analysis of data from the phase III programme. Lupus Sci Med. 2021 Feb;8(1):e000459. doi: 10.1136/lupus-2020-000459. PMID 33568389
- [Derived] Gomez A, Hani Butrus F, Johansson P, Akerstrom E, Soukka S, Emamikia S, Enman Y, Pettersson S, Parodis I. Impact of overweight and obesity on patient-reported health-related quality of life in systemic lupus erythematosus. Rheumatology (Oxford). 2021 Mar 2;60(3):1260-1272. doi: 10.1093/rheumatology/keaa453. PMID 32918459
- [Derived] van Vollenhoven RF, Navarra SV, Levy RA, Thomas M, Heath A, Lustine T, Adamkovic A, Fettiplace J, Wang ML, Ji B, Roth D. Long-term safety and limited organ damage in patients with systemic lupus erythematosus treated with belimumab: a Phase III study extension. Rheumatology (Oxford). 2020 Feb 1;59(2):281-291. doi: 10.1093/rheumatology/kez279. PMID 31302695
- [Derived] Furie R, Petri MA, Strand V, Gladman DD, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Clinical, laboratory and health-related quality of life correlates of Systemic Lupus Erythematosus Responder Index response: a post hoc analysis of the phase 3 belimumab trials. Lupus Sci Med. 2014 Jun 26;1(1):e000031. doi: 10.1136/lupus-2014-000031. eCollection 2014. PMID 25396065
- [Derived] Petri MA, van Vollenhoven RF, Buyon J, Levy RA, Navarra SV, Cervera R, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Baseline predictors of systemic lupus erythematosus flares: data from the combined placebo groups in the phase III belimumab trials. Arthritis Rheum. 2013 Aug;65(8):2143-53. doi: 10.1002/art.37995. PMID 23754628
- [Derived] Strand V, Levy RA, Cervera R, Petri MA, Birch H, Freimuth WW, Zhong ZJ, Clarke AE; BLISS-52 and -76 Study Groups. Improvements in health-related quality of life with belimumab, a B-lymphocyte stimulator-specific inhibitor, in patients with autoantibody-positive systemic lupus erythematosus from the randomised controlled BLISS trials. Ann Rheum Dis. 2014 May;73(5):838-44. doi: 10.1136/annrheumdis-2012-202865. Epub 2013 Mar 22. PMID 23524886
- [Derived] Wallace DJ, Navarra S, Petri MA, Gallacher A, Thomas M, Furie R, Levy RA, van Vollenhoven RF, Cooper S, Zhong ZJ, Freimuth W, Cervera R; BLISS-52 and -76, and LBSL02 Study Groups. Safety profile of belimumab: pooled data from placebo-controlled phase 2 and 3 studies in patients with systemic lupus erythematosus. Lupus. 2013 Feb;22(2):144-54. doi: 10.1177/0961203312469259. Epub 2012 Dec 4. PMID 23213069
- [Derived] van Vollenhoven RF, Petri MA, Cervera R, Roth DA, Ji BN, Kleoudis CS, Zhong ZJ, Freimuth W. Belimumab in the treatment of systemic lupus erythematosus: high disease activity predictors of response. Ann Rheum Dis. 2012 Aug;71(8):1343-9. doi: 10.1136/annrheumdis-2011-200937. Epub 2012 Feb 15. PMID 22337213
- [Derived] Stohl W, Hiepe F, Latinis KM, Thomas M, Scheinberg MA, Clarke A, Aranow C, Wellborne FR, Abud-Mendoza C, Hough DR, Pineda L, Migone TS, Zhong ZJ, Freimuth WW, Chatham WW; BLISS-52 Study Group; BLISS-76 Study Group. Belimumab reduces autoantibodies, normalizes low complement levels, and reduces select B cell populations in patients with systemic lupus erythematosus. Arthritis Rheum. 2012 Jul;64(7):2328-37. doi: 10.1002/art.34400. PMID 22275291
- [Derived] Navarra SV, Guzman RM, Gallacher AE, Hall S, Levy RA, Jimenez RE, Li EK, Thomas M, Kim HY, Leon MG, Tanasescu C, Nasonov E, Lan JL, Pineda L, Zhong ZJ, Freimuth W, Petri MA; BLISS-52 Study Group. Efficacy and safety of belimumab in patients with active systemic lupus erythematosus: a randomised, placebo-controlled, phase 3 trial. Lancet. 2011 Feb 26;377(9767):721-31. doi: 10.1016/S0140-6736(10)61354-2. Epub 2011 Feb 4. PMID 21296403
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HGS1006-C1057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through 48 weeks.
- Belimumab 1 mg/kg: Belimumab 1 mg/kg IV plus standard therapy; belimumab 1 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 48 weeks.
- Belimumab 10 mg/kg: Belimumab 10 mg/kg IV plus standard therapy; belimumab 10 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Started | 287 | 288 | 290
Completed | 226 | 240 | 241
Not Completed | 61 | 48 | 49
Not completed — Withdrawal by Subject | 7 | 6 | 3
Not completed — Adverse Event | 19 | 16 | 15
Not completed — Lack of Efficacy | 16 | 12 | 12
Not completed — Lack of Compliance | 1 | 1 | 1
Not completed — Lost to Follow-up | 4 | 6 | 3
Not completed — Protocol Violation | 7 | 2 | 3
Not completed — Physician Decision | 3 | 2 | 3
Not completed — Other | 4 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 287 | 288 | 290 | 865
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.8) | 35.0 (10.6) | 35.4 (10.8) | 35.5 (11.1)
Age, Customized [Number; unit: participants]
  ≤ 45 years | 225 | 236 | 236 | 697
  Between 45 and 65 years | 57 | 48 | 52 | 157
  ≥ 65 years | 5 | 4 | 2 | 11
Gender [Count of Participants; unit: Participants]
  Female | 270 | 271 | 280 | 821
  Male | 17 | 17 | 10 | 44
Region of Enrollment [Number; unit: participants]
  Europe | 33 | 34 | 31 | 98
  South America | 145 | 143 | 140 | 428
  Southeast Asia | 103 | 106 | 115 | 324
  Australia | 6 | 5 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: SLE Responder Index (SRI) Response Rate at Week 52
Description: Percentage of subjects with a ≥ 4 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
  SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. PGA is a visual analog scale scored from 0 to 3 (1=mild, 2=moderate, 3=severe). BILAG uses a single score for each of the 8 organ domains; range is from severe to no disease (A to E).
Time Frame: Baseline, 52 weeks
Population: Analysis was performed on a modified intention-to-treat (MITT) population, defined as all subjects who were randomized and received at least 1 dose of study agent. Subjects who required rescue SLE medications were declared nonresponders, as were subjects who dropped out or were missing Week 52 data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 287 | 288 | 290
Percentage of participants | 43.6 | 51.4 | 57.6
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0006, Regression, Logistic — For the primary analysis of the primary efficacy endpoint, a step-down sequential testing procedure was used to control the type 1 error; Adjusted for baseline stratification factors (SELENA SLEDAI Score: ≤9 vs ≥10; proteinuria: <2g vs ≥2g per 24hr; Race: African/indig-American vs Other); Odds Ratio (OR) = 1.83, 95% CI [1.30 to 2.59]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.0129, Regression, Logistic — After superiority of 10 mg/kg vs placebo was established, the 1 mg/kg group was tested vs placebo (2-sided alpha=0.05); Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.10 to 2.19]

2. Secondary Outcome: Percent of Subjects With a ≥ 4 Point Reduction From Baseline in SELENA SLEDAI Score at Wk 52.
Time Frame: Baseline, 52 weeks
Population: Analysis was performed on a MITT population, defined as all subjects who were randomized and received at least 1 dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 287 | 288 | 290
Percentage of participants | 46.0 | 53.1 | 58.3
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0024, Regression, Logistic; Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.21 to 2.41]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.0189, Regression, Logistic; Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.07 to 2.14]

3. Secondary Outcome: Mean Change in Physician's Global Assessment (PGA) at Wk 24.
Description: The PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Scores on a 3-point scale
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 287 | 288 | 290
Scores on a 3-point scale | -0.39 (0.03) | -0.44 (0.03) | -0.54 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Adjusted for baseline PGA score and baseline stratification factors
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.2712, ANCOVA; Adjusted for baseline PGA score and baseline stratification factors

4. Secondary Outcome: Mean Change From Baseline in Medical Outcomes 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score (PCS) at Wk 24.
Description: The SF-36 is a generic health related quality of life (HRQOL) measurement. The survey includes 36 questions grouped to 8 domains and 2 summary measures (physical and mental health component, PCS and MCS, respectively) assessing HRQOL. Responses are scored according to the SF-36v2™ manual. A score is calculated for each SF-36 domain based on the patient's response to each question within it. This is then transformed to a scale ranging from 0 (worst) to 100 (best) points. The PCS is norm-based where the mean=50 and standard deviation (SD)=10. Higher scores represent better physical health.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 287 | 288 | 290
Scores on a scale | 3.64 (0.42) | 3.65 (0.43) | 3.58 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.8870, ANCOVA; Adjusted for the baseline PCS score and baseline stratification factors
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.8127, ANCOVA; Adjusted for the baseline PCS score and baseline stratification factors

5. Secondary Outcome: Percent of Subjects Whose Average Prednisone Dose Has Been Reduced by ≥ 25% From Baseline to ≤ 7.5 mg/Day During Weeks 40 Through 52
Time Frame: Baseline, Weeks 40 through 52
Population: Analysis was performed on a MITT population, defined as all subjects who were randomized and received at least 1 dose of study agent. Includes only subjects with baseline prednisone dose > 7.5 mg/day
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 192 | 204 | 204
Percentage of participants | 12.0 [0 to 0] | 20.6 [1.08 to 3.31] | 18.6 [0.99 to 3.08]
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0526, Regression, Logistic; Adjusted for baseline prednisone dose level and baseline stratification factors; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.99 to 3.08]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.0252, Regression, Logistic; Adjusted for baseline prednisone dose level and baseline stratification factors; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.08 to 3.31]

6. Other Pre Specified Outcome: Adverse Events (AE) Overview
Description: SEE ALSO ADVERSE EVENTS RESULTS SECTION
Time Frame: Up to 56 Weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 287 | 288 | 290
Percentage of participants
  Percent of patients with at least 1 AE | 91.6 | 91.7 | 91.7
  Percent of patients with at least 1 Serious AE | 12.5 | 16.3 | 14.1
  Percent of patients with an AE resulting in death | 1.0 | 0.7 | 1.4

ADVERSE EVENTS:
Time Frame: Up to 56 weeks.
Description: Includes AEs reported in subjects from first dose of study agent throughout the study up to the Week 52/Exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (HGS 1006-C1074/NCT00712933).
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 36/287 | 47/288 | 41/290
Other Adverse Events (participants affected / at risk) | 222/287 | 219/288 | 223/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=287) | Belimumab 1 mg/kg (N=288) | Belimumab 10 mg/kg (N=290)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Pericarditis lupus (Cardiac disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Ocular vasculitis (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Lupus enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 1
Vasculitis gastrointestinal (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Infusion related reaction (General disorders) | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 4
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 4 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Ecthyma (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 2 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 1
Herpes zoster multi-dermatomal (Infections and infestations) | 0 | 2 | 0
Joint abscess (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 2
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Phlebitis infective (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 4 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 3
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 1
Personality disorder (Psychiatric disorders) | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 3 | 3
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 2 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=287) | Belimumab 1 mg/kg (N=288) | Belimumab 10 mg/kg (N=290)
Anaemia (Blood and lymphatic system disorders) | 13 | 13 | 15
Abdominal pain upper (Gastrointestinal disorders) | 18 | 8 | 13
Diarrhoea (Gastrointestinal disorders) | 19 | 28 | 30
Dyspepsia (Gastrointestinal disorders) | 15 | 11 | 11
Gastritis (Gastrointestinal disorders) | 7 | 10 | 15
Mouth ulceration (Gastrointestinal disorders) | 18 | 5 | 12
Nausea (Gastrointestinal disorders) | 31 | 16 | 23
Vomiting (Gastrointestinal disorders) | 13 | 16 | 14
Fatigue (General disorders) | 12 | 17 | 18
Oedema peripheral (General disorders) | 21 | 20 | 17
Pyrexia (General disorders) | 17 | 15 | 16
Bronchitis (Infections and infestations) | 7 | 21 | 16
Cystitis (Infections and infestations) | 9 | 12 | 22
Gastroenteritis (Infections and infestations) | 16 | 20 | 12
Influenza (Infections and infestations) | 25 | 22 | 33
Nasopharyngitis (Infections and infestations) | 23 | 30 | 20
Pharyngitis (Infections and infestations) | 7 | 16 | 15
Upper respiratory tract infection (Infections and infestations) | 47 | 41 | 36
Urinary tract infection (Infections and infestations) | 24 | 27 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 21 | 32
Arthritis (Musculoskeletal and connective tissue disorders) | 18 | 13 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 25 | 19
Dizziness (Nervous system disorders) | 23 | 16 | 15
Headache (Nervous system disorders) | 75 | 58 | 66
Insomnia (Psychiatric disorders) | 14 | 9 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 23 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 10 | 17
Hypertension (Vascular disorders) | 30 | 24 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center trials, no investigator will be authorized to publish study results from an individual center until the earlier of the multi-center trial results are published or 12 months after the end or termination of the multi-center trial at all sites. All manuscripts and abstracts must be submitted to the sponsor for review at least 30 days prior to submission for publication or for presentation at a scientific meeting. The sponsor may delay publication for up to 3 months.